CLINICAL TRIAL: NCT04347850
Title: A Cohort of Patients With Possible or Confirmed SARS-CoV-2 (COVID-19) Infection, From Diagnosis to Long-term Follow-up
Brief Title: A Cohort of Patients With Possible or Confirmed SARS-CoV-2 (COVID-19)
Acronym: COVIDothèque
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0185
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: SARS-CoV-2; COVID-19
Keywords: presence of COVID-19 symptoms; COVID-19 infection
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, total blood, urine, stool, oral fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient with Covid-19 confirmed (middle form): Covid-19 confirmed: middle form
  Interventions: Other: blood sample
- Patient with Covid-19 confirmed (severe form): Covid-19 confirmed : severe form
  Interventions: Other: blood sample
- Patient with Covid-19 not confirmed: Covid-19 not confirmed
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — Collection

SUMMARY:
SARV-CoV-2 infection was considered pandemic on March 11, 2020. The SARV-CoV-2 epidemic affected France from the beginning of March, spreading in particular from a 4-day large evangelical meeting of 2500 people on February 17 in the city of Mulhouse (North East of France). The Montpellier University Hospital has set up a clinical pathway for people suspected of being infected with SARV-CoV-2 because of signs compatible with pneumonia (screening criteria in France during the study period). This includes an emergency department, an infectious disease department dedicated to the surveillance of infected people requiring hospital treatment, and an intensive care unit for the most severe cases. The diagnosis of infection with SARV-CoV-2 was confirmed in approximately 20% of people initially referred in this special care system.

The main objective of this cohorte is the collection of clinical data and biological samples from care for non-interventional research on the patients with a possible or confirmed SARS-CoV -2 infection, from diagnosis to long-term follow-up.

ELIGIBILITY:
Inclusion criteria:

- Patients care at the Montpellier University Hospital suspected of a COVID-19 infection

Exclusion criteria:

* Patient opposed to the use of his data for research purposes
* Patient deprived of liberty by judicial decision
* Patient not affiliated to a social security scheme

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a possible or confirmed SARS-CoV -2 infection, from diagnosis to long-term follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of confirmed COVID-19 | 1 day
  Number of confirmed COVID-19

SECONDARY OUTCOMES:
Number of severe COVID-19 | 1 day
  Number of severe COVID-19
Identification and validation of predictive biomarkers of a poorer respiratory evolution associated with positive testing for SARS-CoV-2 infection | 1 day
  CORO-TRI substudy
Evaluate the morbidity and mortality and these risk factors linked to Covid-19 in the congenital heart disease population in France | 1 day
  COVID-CHD substudy
Identify the characteristics of physiotherapy care for patients with COVID-19 in intensive care | 1 day
  Physio-Covid substudy
To assess the accuracy and prognostic performance of clinical and biological parameters measured on admission to the emergency department to stratify patients suspected of COVID-19 | 1 day
  Covida substudy
Evaluate diagnostic tests for olfactory function in relation to the RT-PCR procedure | 1 day
  Olfa-covid substudy
Assessment of Extra Vascular Lung Water and Pulmonary Permeability by transpulmonary thermodilution in critically ill patients with Coronavirus Disease 2019 pneumonia under invasive mechanical ventilation | 1 day
  PiCCOVID substudy
Description of trans pulmonary motor pressure in COVID 19+ patients in severe stage in intensive care | 1 day
  TRANSPULMONARY-COVID19 substudy
Immuno-monitoring of COVID-19 positive patients | 1 day
  CytoCOVID substudy
Characterization in clinical proteomics of the SARS-CoV-2 spike protein | 1 day
  ProteoCOVID substudy
Diagnosis of endocrine dysfunctions in Covid-19 | 1 day
  Dyhor-19 substudy
describe the occurrence of Covid19 infection in patients with systemic lupus erythematosus treated with hydroxychloroquine over the long term | 1 day
  Lupus substudy
Acral cutaneous thrombotic vasculopathy and Covid-19 infection : search for acquired thrombophilia and interferon-alpha signature | 1 day
  Vasculopathy substudy
Evaluation of a COVID-19 screening strategy combining chest low dose CT and RT-PCR test for patients admitted for surgical or interventional procedures during the COVID 19 outbreak | 1 day
  COVID-Scan study

CONTACTS AND LOCATIONS:
Overall Officials: Edouard TUAILLON, MD; PhD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No
NC

REFERENCES:
- [Derived] Capelli N, Domitien Payet L, Alcocer Cordellat C, Pisoni A, Engelmann I, Van de Perre P, Jeziorski E, Tuaillon E. SARS-CoV-2 nucleocapsid antigen in plasma of children hospitalized for COVID-19 or with incidental detection of SARS-CoV-2 infection. J Med Virol. 2024 Jan;96(1):e29358. doi: 10.1002/jmv.29358. PMID 38180230